CLINICAL TRIAL: NCT03628001
Title: A Prospective, Randomized, Multicenter Study Comparing Sems Placement With and and Without Biliary Sphincterectomy in Patients With Malignant Biliary Obstruction (ES vs noES-1)
Brief Title: A Study Comparing Sems Placement With and and Without Biliary Sphincterectomy in Patients With Malignant Biliary Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1442
Record Dates: First submitted 2018-04-03; First posted 2018-08-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Bile Duct Obstruction
Keywords: Endoscopic retrograde cholangiopancreatography (ERCP); Distal malignant bile duct obstruction; Sphincterotomy
MeSH Terms: conditions — Cholestasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Other): ERCP with (Group A) ES before biliary SEMS placement
  Interventions: Procedure: ERCP
- B (Other): ERCP without (Group B) ES before biliary SEMS placement
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Pts will be randomized with or without sphinterectomy.

SUMMARY:
Background and rationale Placement of biliary self expanding metal stent (SEMS) is indicated when malignant common bile duct obstruction is encountered.

Currently, there is still controversy regarding the use of endoscopic sphincterotomy (EST) before the placement of biliary stents. EST may facilitate insertion of self expandable metal stent (SEMS) and also help avert the development of pancreatitis from stent-related occlusion of the pancreatic duct. On the other hand, ES is also independently associated with pancreatitis, bleeding, and perforation.

Latest European guidelines indicate that EST is not necessary for inserting single plastic or metal biliary stents, nevertheless a more recent meta analysis showed that ES may decrease the rate of PEP.

Population and patient selection criteria All the patient referred for endoscopic retrograde cholangiopancreatography (ERCP) due to malignant bile duct obstruction.

Study design and study duration Prospective randomized, multicenter study. 18 months.

Description of study treatment/product/intervention All the patients will be randomly assigned to undergo ERCP with (Group A) or without (Group B) ES before biliary SEMS placement.

All the endoscopic procedures will be performed by experienced endoscopist in the endoscopy suite.

All the procedure will be conducted under deep sedation. SEMS placed will be fully covered.

Objectives To assess the need for EST before SEMS placement in patients with malignant bile duct obstruction.

To evaluate immediate (periprocedural) and delayed (30 days) post ERCP complications including pancreatitis, SEMS migration, bleeding and perforation.

Statistical methods, data analysis A sample size analysis to detect superiority at 5% significance level and a power of 80% showed that 500 patients had to be enrolled in each group.

Continuous variables such age will be reported in terms of their mean and range, and t-test will be done to test their main difference.

X square test or Fisher exact test will be carried out for statistical analysis to compare rates of total complications between the two groups and rates of pancreatitis, bleeding, stent migration and perforation.

Wilcoxon Mann-Withney test will be used for comparison of means between 2 continuous variables. A single-tailed P value of less than 0,05 is considered significant.

Study time table Project starting date: 15-7-2015 Project completion of patients accrual: 15-10-2016 Project completion of data collection: 15-11-2016 Project data analysis: 15-2-2017 Project presentation of scientific report: 15-4-2017

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for endoscopic retrograde cholangiopancreatography
* Malignant bile duct obstruction
* Signed written informed consent
* Age > 18

Exclusion Criteria:

* Inability to provide inform consent
* Pregnancy or lactation
* Suspected perforation of the GI tract
* Anatomical alterations due to previous surgery (Billroth surgery)
* Coagulation alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and type of complications after ERCP. | 18 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Gastroenterology Department, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT03628001/Prot_SAP_000.pdf